CLINICAL TRIAL: NCT02232659
Title: SynCardia 70cc Temporary Total Artificial Heart (TAH-t) for Destination Therapy (DT)
Brief Title: SynCardia 70cc TAH-t for Destination Therapy (DT)
Acronym: RA-540
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SynCardia Systems. LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SynCardia 70cc TAH-t for DT
Record Dates: First submitted 2014-09-02; First posted 2014-09-05 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Life-threatening; Biventricular Heart Failure; Ineligible for Cardiac Transplant
Keywords: SynCardia; Total Artificial Heart; Biventricular heart failure; Ineligible for cardiac transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primary Arm (Experimental): Use of the SynCardia 70cc TAH-t for Destination Therapy to support an HDE Application.
  Interventions: Device: 70cc TAH-t for Destination Therapy
- Secondary Arm (Experimental): Use of the SynCardia 70cc TAH-t for Destination Therapy in a less-restrictive patient population to further characterize the use of the 70cc TAH-t for DT.
  Interventions: Device: 70cc TAH-t for Destination Therapy

INTERVENTIONS:
Device: 70cc TAH-t for Destination Therapy — Use of the approved SynCardia 70cc TAH-t for patients who are in biventricular failure (approved use), but who are ineligible for cardiac transplant (experimental use).

SUMMARY:
The SynCardia 70cc temporary Total Artificial Heart (TAH-t) is approved by the U.S. Food and Drug Administration (FDA) for use as a bridge to transplant for patients at risk of imminent (about to happen) death from irreversible biventricular heart failure.

The purpose of this research study is to evaluate whether the TAH-t can support patients with life-threatening irreversible biventricular heart failure who are not eligible for transplantation. The TAH-t, when used for patients who are not eligible for transplant, is considered to be an investigational (not approved by FDA) use. This use is called destination therapy (DT).

Nineteen (19) patients with life-threatening, biventricular failure who are not eligible for cardiac transplant will be enrolled in the Primary Arm of the study and followed for up to six months post-TAH-t implant. Safety will be evaluated by reviewing the adverse events that are experienced by the enrolled subjects and comparing them to previous experience of TAH-t patients who were waiting for a heart transplant. Since approximately 74% of patients with this condition would not be expected to live beyond six months, the benefit of the TAH-t for DT will be confirmed based on survival to six months without experiencing permanent disabling stroke-related deficits. After the six month follow-up visit, patients will continue to be followed under the study for up to five (5) years postTAH-t implant [every six months for up to two years while supported with the TAH-t implant and then annually for another three years].

Up to an additional 19 patients may be enrolled in the Secondary Arm of the study to further characterize the use of the TAH-t for DT in a broader patient population. Follow-up would be the same for patients enrolled in both arms of the study.

DETAILED DESCRIPTION:
On 15 October 2004, the SynCardia temporary Total Artificial Heart (TAH-t) received Food and Drug Administration (FDA) approval (Premarket Approval Application [PMA] #P030011) for in-hospital use as a bridge to transplant (BTT) in cardiac transplant-eligible candidates at risk of imminent death from biventricular failure.

On 2 March 2012, FDA granted a Humanitarian Use Designation (HUD) to the 70cc TAH-t System for use as Destination Therapy (DT) in patients at risk of imminent death from irreversible biventricular heart failure who are not eligible for transplant and have a body surface area (BSA) >1.7m. This clinical study is intended to determine the safety and probable benefit of the 70cc TAH-t for use in DT and support a Humanitarian Device Exemption (HDE) application for this new indication for the TAH-t System.

The SynCardia TAH-t System is a pulsatile biventricular device that replaces a patient's native ventricles and valves by pumping blood to both the pulmonary and systemic circulation.

The TAH-t System for DT consists of the implantable TAH-t with SynHall Valves, powered by PMA-approved external pneumatic drivers [the Circulatory Support System (CSS) Console, the Companion 2 Driver System and the Freedom Driver System]. The TAH-t System is intended to be implanted in the operating room by a qualified surgeon and is capable of supporting the patients both inside and outside the hospital.

The SynCardia TAH-t for DT is indicated for refractory advanced heart failure patients with biventricular failure who are not candidates for cardiac transplant because of the presence of contraindications to transplant, including cancer, advanced age, obesity, end-stage diabetes mellitus, high panel reactive antibodies (PRAs), non-cardiac congenital defects, contraindications to immunosuppression, lack of social support, poor medical compliance, neurological impairment or other co-morbidities with a poor prognosis for survival. Patients with life-threatening, irreversible biventricular failure who are not eligible for transplant currently have no alternative but death.

The rationale for conducting this study is based on the results of clinical studies in the bridge-to-transplant (BTT) patient population, together with the in vitro design verification and validation testing, in vitro reliability testing, and clinical reliability experience of more than thirty years.

The study design is a prospective, non-randomized, two-treatment arm, multi-center study. Nineteen (19) patients will be enrolled in the Primary Arm at up to 30 investigational sites to support an HDE for the use of the TAH-t as DT. Up to an additional 19 patients may be enrolled in the Secondary Arm to futher characterize the use of the TAH-t for DT in a broader patient population.

Patients treated with the 70cc TAH-t System for DT under the Primary Arm will be adult male and female patients between the ages of 19 and 75 years old with a BSA ≥1.7m2 with life-threatening irreversible biventricular failure who are not eligible for a heart transplant (as determined by the implanting center at the time of implant assessment) and who meet the enrollment criteria defined in the clinical protocol. Patients treated with the 70cc TAH-t System for DT under the Secondary Arm will be adult male and female patients who are at least 19 years old, are not eligible for a heart transplant (as determined by the implanting center at the time of implant assessment), and who meet the less restrictive enrollment criteria defined in the clinical protocol.

The risks to which the TAH-t subjects will be exposed in this clinical investigation are expected to be no more than the well-characterized risks of the PMA-approved TAH-t System when used for the bridge-to-transplant population and have been mitigated by the design and testing of the TAH-t System.

The primary objective of the SynCardia temporary Total Artificial Heart (TAH-t) for DT Study is to evaluate whether the TAH-t can support patients with life-threatening irreversible biventricular heart failure who are ineligible for cardiac transplantation (as determined by the implanting center at time of implant screening assessment), without experiencing permanent disabling stroke-related deficits (as evidenced by a Modified Rankin Scale score of 0 - 2). The other primary objective of the study is to evaluate whether the safety profile of the device, when used for DT, is acceptable.

Probable benefit is defined as survival to six months on TAH-t System support with the same implanted TAH-t, without experiencing permanent disabling stroke-related deficits. This patient population, without treatment, has a poor prognosis of survival. Per M.L.A. Haeck, "Patients with drug refractory end-stage HF [heart failure] receiving support with inotropic drugs [have] a 3-, 6-, and 12-month survival of 51%, 26%, and 6%, respectively, with a mean survival of only 3.4 months."1

The study success criteria are: alive on the original TAH-t and free from permanent disabling stroke-related deficits (as evidenced by Modified Rankin Scale score of 0 - 2) at six months post-implant (or transplanted prior to six months post-implant). For the study to be considered a success, eight of the 19 subjects either must be alive at six months on the original TAH-t implant, without experiencing a permanent disabling stroke deficit, or have become transplant eligible (or have been transplanted).

The safety endpoints will be captured according to the Intermacs Registry AE definitions and will be assessed according to the same data collection schedule followed under the Intermacs Registry protocol. Secondary safety endpoints will be the incidences of major infection (sepsis), neurological events (ischemic or hemorrhagic cardiovascular accident [CVA]), chronic renal dysfunction, and the rate of major device failures/malfunctions, each defined per the Intermacs definitions. A performance goal for each has been established based on the previous experience of TAH-t patients who were waiting for a heart transplant.

All subjects will be followed in the study from the date of TAH-t implant until six months post-implant, cardiac transplantation, death, or withdrawal from study, whichever occurs first. Data from the six month post-TAH-t implant period will be used to support an HDE application. After the six month follow-up visit, patients will continue to be followed under the study for up to five (5) years post-TAH-t implant [every six months for up to two years while supported with the TAH-t implant and then annually for another three years].

1 Neth Heart J (2012) 20:167-175 15 November 2011

ELIGIBILITY:
Primary Arm

Inclusion Criteria:

1. Patients with ife-threatening, irreversible biventricular heart failure (Intermacs Patient Profile Classifications 1 - 4)
2. Ineligible for cardiac transplantation (e.g., contraindication to immunosuppression, cancer, elevated panel reactive antibodies [PRAs]) as determined by the implanting center at time of implant screening assessment.
3. On optimal medical management and failing to respond or failing DT VAD therapy (continuing to decline)
4. Ambulatory without assistance
5. Patients between 19 and 75 years of age
6. Patients with Body Surface Area (BSA) of ≥ 1.7m2
7. Sternum to T10 distance > 10cm OR adequate room in chest as determined by 3-D imaging assessment or by other standard clinical assessments

Exclusion Criteria:

1. Cardiac transplant-eligible patients
2. Patients who cannot be adequately anticoagulated on the TAH-t
3. Patients with insufficient space in the chest
4. Patients on ECMO support
5. Patients with Cirrhosis (evidenced by ultrasound, CT scan, or positive biopsy)
6. Patients with Acute or Chronic Renal dysfunction (per Intermacs AE Definitions)
7. Patients with cardiac cachexia (e.g., pre-albumin <17, fragility, and catabolic/anabolic imbalance)
8. Patients with a comorbidity that has a poor prognosis of survival beyond six months
9. Patients with insufficient social support or who have demonstrated non-compliance with medical instructions (as determined by the Principal Investigator)

Secondary Arm

Inclusion Criteria:

1. Patients who are NOT eligible to participate in the Primary Arm
2. Patients with life-threatening, irreversible biventricular heart failure (Intermacs Patient Profile Classifications 1 - 7)
3. Ineligible for cardiac transplantation (as determined by the implanting center at time of implant screening assessment).
4. On optimal medical management and failing to respond or failing DT VAD therapy (continuing to decline)
5. Patients 19 years of age or older
6. Sternum to T10 distance > 10cm OR adequate room in chest as determined by 3-D imaging assessment or by other standard clinical assessments

Exclusion Criteria:

1. Patients who are less than 19 years old
2. Cardiac transplant-eligible patients
3. Patients with Cirrhosis (evidenced by ultrasound, CT scan, or positive biopsy)
4. Patients with Chronic Renal dysfunction (per Intermacs AE Definitions)
5. Patients with insufficient space in the chest
6. Patients who cannot be adequately anticoagulated on the TAH-t
7. Patients with insufficient social support or who have demonstrated non-compliance with medical instructions (as determined by the Principal Investigator)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Probable Benefit | Six Months
  Alive on original TAH-t and free from permanent disabling stroke-related deficits (as evidenced by Modified Rankin Scale score of 0 - 2) at six months post-implant (or transplanted prior to six months post-implant).

SECONDARY OUTCOMES:
Safety | Six Months
  Adverse Events (AEs) will be captured according to the Intermacs Registry AE definitions and will be assessed according to the same data collection schedule followed under the Intermacs Registry protocol for up to two years post-implant. In addition to reporting of rate, number and percent of subjects experiencing each adverse event, individual performance goals have been determined for four adverse event categories, based on the previous experience of patients supported by the TAH-t while awaiting cardiac transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Copeland, MD, Principal Investigator
Locations (7):
- United States (7):
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Memorial Hermann Hospital, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin